CLINICAL TRIAL: NCT05024487
Title: Risk Level Determination of Vascular Complications Due to Autonomic Dysreflexia in Spinal Cord Injured Individuals
Brief Title: Prevention of Complications Due to Autonomic Dysreflexia in SCI Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assoc. Prof. Jiri Kriz, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Assoc. Prof. Jiri Kriz, MD, PhD, Clinical Professor, University Hospital, Motol
Organization: University Hospital, Motol (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCI_DYSREFLEXIA_2021
Record Dates: First submitted 2021-08-13; First posted 2021-08-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Autonomic Dysreflexia; Spinal Cord Injuries
Keywords: Autonomic Nervous System; Spinal Cord Injury; Prevention
MeSH Terms: conditions — Autonomic Dysreflexia; Spinal Cord Injuries | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The correlation between blood pressure level, dermal resistance level, and subjective symptoms caused by triggered AD below the level of the lesion will be performed in a group of SCI people.
  Interventions: Diagnostic Test: Clinical Examination

INTERVENTIONS:
Diagnostic Test: Clinical Examination — Given the most frequent causes of AD, the above-mentioned trigger stimuli will be used. All these procedures are commonly used in SCI people.
  Other Names: Pinprick in sacral dermatome 4/5 (a part of International Standards for Neurological Classification of Spinal Cord Injury - ISNCSCI); Deep Anal Pressure (a part of ISNCSCI); Intermittent catheterization of the bladder; In absence of one of above-mentioned stimuli, stretching of hamstrings during elevation of legs will be performed

SUMMARY:
Autonomic dysreflexia (AD) is a syndrome of unbalanced response of the sympathetic system to noxious stimuli below the level of spinal cord injury (SCI), characterized by paroxysmal hypertension. Mostly, it is combined with symptoms such as pounding headache, slowed heart rate, and upper body flushing, but it can also be asymptomatic. When resulting in hypertensive crisis, it can be life-threatening and result in seizures, cardiac arrest, retinal or subarachnoid hemorrhages, stroke, and even death.

The aim of this study is to determine the risk level of vascular complications in SCI people by correlating the clinical symptoms with their individual perception during AD triggered below the level of injury.

DETAILED DESCRIPTION:
After spinal cord injury, the disruption of descending vasomotor pathways to sympathetic neurons causes their hyperexcitability. When irritated by noxious stimuli below the level of injury, a massive sympathetic reflex is triggered, causing widespread vasoconstriction. If the neurological level of injury is at or above T6, this vasoconstriction can lead to progressive hypertension possibly involving the splanchnic vessels.

In response to hypertension, the baroreflex system lowers blood pressure by reducing heart rate and decreasing the activity of sympathetic neurons. However, a decrease in peripheral vascular resistance below the injury level does not occur because of the disruption of descending vasomotor pathways to sympathetic neurons. Thus, hypertension persists until the triggering stimulus is removed. Hypertensive crises can result in vascular complications like cardiac arrest, retinal or subarachnoid hemorrhages, stroke, and even death. Vasodilatation above the lesion level is accompanied by characteristic signs and symptoms such as upper body flushing and sweating, and a pounding headache. Sometimes bradyarrhythmia, seizures, nausea, or anxiety can occur. Unfortunately, AD can take place asymptomatically in almost 40 %. These asymptomatic individuals are at high risk of life-threatening complications mentioned above.

The most frequent AD triggers are overfilled bladder or bowel. Nevertheless, it can be any irritating stimuli below the level of injury, i.e., skin lacerations, ingrown toenails, or pressure sores.

Higher intensity of perception of clinical symptoms accompanying AD decreases the risk of vascular complications. People who perceive subjective signs of AD even in slightly elevated blood pressure can eliminate irritating stimuli or use an antihypertensive medication and thus avoid life-threatening complications. On contrary, people who cannot perceive the signs intensely enough are at a significantly higher risk of vascular complications.

The aim of this study is to determine the risk level of vascular complications in SCI people. The AD will be triggered below the injury level so that the clinical symptoms can be correlated with their subjective individual perception. Moreover, the development of a method allowing capturing AD episodes in individuals without subjective signs is intended.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old female and male patients
* People in chronic phase (more than 12 months) after traumatic or ischemic spinal cord lesion
* People with Neurological Level of Injury C3-T6 and ASIA Impairment Scale A-B according to ISNCSCI
* Written informed consent

Exclusion Criteria:

* People with acute infection or other suddenly incurred complication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure monitoring | During the intervention
  Continuous blood pressure and heart rate monitoring will be recorded using Finapres device.
  The risk level will be determined according to the value of systolic blood pressure (SBP):
  1. Low risk - SBP to 150 mmHg
  2. Moderate risk - SBP 150-200 mmHg
  3. High risk - SBP above 200 mmHg

SECONDARY OUTCOMES:
Dermal sweating | During the intervention
  Wrist sweating will be monitored using a measure of dermal resistance with range 0-5 MΩ (difference 0,1 kΩ, accuracy 0,15 %) and 5-32 MΩ (difference 10 kΩ, accuracy 1 %) and sampling frequency 10 second.
  Regarding the AD symptoms, level of dermal resistance decrease corresponds to increase of sweating.
Assessment of symptoms | During the intervention
  Subjective individual symptoms are divided into three groups, according to their severity (minimum value: mild symptoms, maximum: strong symptoms):
  1. Mild symptoms - shivers on the nape or on the back
  2. Moderate symptoms - sweating on the forehead, neck or upper extremities
  3. Strong symptoms - pounding headache, nausea
ADFSCI questionnaire | During the intervention
  The ADFSCI (Autonomic Dysfunction Following Spinal Cord Injury) questionnaire provides information about individual symptoms of blood pressure (BP) instability. The ADFSCI is a 24-item questionnaire consisting of four parts: demographics, medication, AD, and hypotension. The AD and hypotension parts include 10 and 7 items, respectively, each using a 5-point scale to score the frequency and severity of hyper- or hypotensive symptoms with a range of 0 ∼ 204 (highest BP instability) points.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Kriz, MD, PhD, Principal Investigator — Spinal Cord Unit, University Hospital Motol
Locations (1):
- Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Machac S, Radvansky J, Kolar P, Kriz J. Cardiovascular response to peak voluntary exercise in males with cervical spinal cord injury. J Spinal Cord Med. 2016 Jul;39(4):412-20. doi: 10.1080/10790268.2015.1126939. Epub 2015 Dec 28. PMID 26707873
- [Background] Kriz J, Andel R, Hakova R. Delayed diagnosis of an unsuspected pelvic fracture in a patient with tetraplegia. J Spinal Cord Med. 2014 Jul;37(4):425-8. doi: 10.1179/2045772313Y.0000000178. Epub 2014 Jan 3. PMID 24621047
- [Background] Kriz J, Relichova Z. Intermittent self-catheterization in tetraplegic patients: a 6-year experience gained in the spinal cord unit in Prague. Spinal Cord. 2014 Feb;52(2):163-6. doi: 10.1038/sc.2013.154. Epub 2013 Dec 17. PMID 24343054